CLINICAL TRIAL: NCT06525636
Title: A Multicenter, Open-label, Phase 1/2, Dose-escalation and Subsequent Safety Extension Study of Subcutaneous KK8123 in Adult Patients With X-linked Hypophosphatemia
Brief Title: A First-in-human Study of KK8123 in Adults With X-linked Hypophosphatemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8123-001
Record Dates: First submitted 2024-05-10; First posted 2024-07-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: X-linked Hypophosphatemia
Keywords: Gene Mutation; Bone Disease; Metabolic Disease; Musculoskeletal Disease,; Rare Disease; Hypophosphatemia; Familial Renal Tubular Transport; Inborn Errors; Kidney Diseases
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Bone Diseases; Metabolic Diseases; Musculoskeletal Diseases; Rare Diseases; Hypophosphatemia; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part I: Cohort 1 (Experimental): Low Dose, single dose of KK8123
  Interventions: Drug: KK8123
- Part I: Cohort 2 (Experimental): Mild dose, multiple doses of KK8123
  Interventions: Drug: KK8123
- Part I: Cohort 3 (Experimental): High dose, multiple doses of KK8123
  Interventions: Drug: KK8123
- Part I: Cohort 4 (Experimental): Optional, multiple doses of KK8123
  Interventions: Drug: KK8123
- Part 2: Extension Period (Experimental): High dose, multiple doses as confirmed for Cohort 3 of KK8123.
  Interventions: Drug: KK8123

INTERVENTIONS:
Drug: KK8123 — Subcutaneous administration

SUMMARY:
A first-in-human study of KK8123 in adults with X-linked hypophosphatemia.

DETAILED DESCRIPTION:
Study 8123-001 is a Phase 1/2, multicenter, open-label, dose-escalation study to assess the safety, tolerability, PK and PD of KK8123, with an optional safety extension period. This study is comprised of a Screening Period followed by Part 1 and Part 2. The Screening Period will last up to 28 days (including obtaining informed consent). Part 1 is a Dose Escalation Period consisting of a nominal (planned) Treatment Period (all cohorts) and Observation Period of 32 to 44 weeks, and Part 2 is an optional Extension Period.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Inclusion Criteria:

  1. Male or female patients aged 18 to 65 years inclusive at the time of signing the ICF.
  2. Body weight is at least 40 kg.
  3. Diagnosed with XLH (as documented by the investigator).
  4. Have a value of fasting serum phosphorus < 2.5 mg/dL (0.81 mmol/L) at Screening.
  5. Have a value of renal TmP/GFR < 2.5 mg/dL (0.81 mmol/L) at Screening.
  6. eGFR ≥ 60 mL/min (using the Chronic Kidney Disease Epidemiology Collaboration equation [Inker, 2021]) at Screening.
  7. Have a corrected serum calcium level < 10.8 mg/dL (2.7 mmol/L) at Screening.
  8. Provide a signed ICF.
  9. Agree not to change diet and exercise regimen from one week prior to dosing to end of study.
  10. Have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study (female participants only).
  11. If taking chronic pain medications (including narcotic pain medications/opioids), must be on a stable regimen for at least 21 days prior to the Screening visit, and be willing to maintain medications at the same stable dose(s) and schedule throughout the clinical trial. The dose must not exceed 60 mg oral morphine equivalents/day.
  12. Be willing to use a method of contraception following local country guidelines while participating in the study and for 5 months after the last dose (all sexually active participants of childbearing potential).

      Women of non-childbearing potential are defined as permanently sterile (i.e., due to tubal ligation at least one year before Screening, hysterectomy or bilateral oophorectomy) or postmenopausal (defined as at least 12 months post cessation of menses without an alternative medical cause).

      Postmenopausal status of female participants will be confirmed with a Screening serum follicle-stimulating hormone level >40 mIU/mL.
  13. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments.

Exclusion Criteria:

* Part 1: Exclusion Criteria:

  1. For XLH patients previously treated with burosumab, use of burosumab within 7 months prior to ICF signature.
  2. Prior history of positive test for human immunodeficiency virus antibody, positive test for hepatitis B surface antigen, and/or hepatitis C virus antibody at Screening.
  3. History of hypersensitivity to any ingredient of any therapeutic monoclonal antibody.
  4. Have an active infection.
  5. Grade 3 or greater nephrocalcinosis as confirmed by renal ultrasound.
  6. Uncontrolled diabetes mellitus at Screening.
  7. History of known immunodeficiency.
  8. History of alcoholism or drug abuse.
  9. History of donation of blood within 60 days prior to Screening.
  10. Use of any IP or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
  11. Use of any therapeutic mAb within 90 days prior to Screening.
  12. Use of pharmacologically active vitamin D, its metabolites or analogs, oral phosphate for treatment of XLH, aluminum hydroxide antacids, acetazolamide, thiazide diuretics, and/or systemic corticosteroids within 14 days prior to Screening. If the participant takes any of these medications, a washout period of 14 days will be required after signing the ICF and before any other screeening assessments begin.
  13. Use of medication to suppress PTH (e.g., calcimimetics) within 2 months prior to Screening and for the duration of the study.
  14. Use of denosumab within 6 months prior to Screening.
  15. Use of oral bisphosphonates in the 2 years prior to Screening.
  16. Use of teriparatide or abaloparatide in the 2 months prior to Screening.
  17. Plasma iPTH ≥ 2.5 × ULN at Screening.
  18. Planned or recommended orthopedic surgery during the study.
  19. History of traumatic fracture or orthopedic surgery within 6 months prior to Screening.
  20. Participants who are lactating.
  21. Current active and symptomatic COVID-19 infection at Day -1.
  22. Presence or history of any condition that, in the view of the investigator, places the participant at high risk of poor treatment compliance or of not completing the study, or that would confound safety or interpretation of results.

Part 2: Inclusion Criteria:

1. Completion of relevant cohort in Part 1 of the study.
2. Provide a signed informed consent after the nature of Part 2 of the study has been explained.
3. Body weight is at least 40 kg.
4. Negative pregnancy test at Week 0 of Part 2 and willing to have additional pregnancy tests until the end of the study (female participants only).
5. If taking chronic pain medications (including narcotic pain medications/opioids), must be on a stable regimen for at least 21 days prior to Week 0 of Part 2, and be willing to maintain medications at the same stable dose(s) and schedule throughout the study. The dose must not exceed 60 mg oral morphine equivalents/day.
6. Be willing to use a method of contraception following local country guidelines while participating in the study and for 5 months after the last dose (all sexually active participants of childbearing potential). Women of non-childbearing potential are defined as permanently sterile (i.e., due to tubal ligation at least one year before Screening, hysterectomy or bilateral oophorectomy) or postmenopausal (defined as at least 12 months post cessation of menses without an alternative medical cause). Postmenopausal status of female participants will be confirmed with a Week 0 serum follicle-stimulating hormone level >40 mIU/mL.
7. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with all the assessments.

Part 2: Exclusion Criteria:

1. Use of burosumab following completion of Part 1 of the study.
2. Have an active infection.
3. Donation of blood within 60 days prior to Week 0 of Part 2.
4. Use of any investigational product other than KK8123, or investigational medical device, within 30 days prior to Week 0 of Part 2, or requirement for any investigational agent prior to completion of all scheduled study assessments.
5. Use of any therapeutic mAb other than KK8123 within 90 days prior to Week 0 of Part 2.
6. Use of pharmacologically active vitamin D, its metabolites or analogs, oral phosphate for treatment of XLH, aluminum hydroxide antacids, acetazolamide, thiazide diuretics, and/or systemic corticosteroids within 14 days prior to Week 0 of Part 2.
7. Use of medication to suppress PTH (e.g., calcimimetics) within 2 months prior to Week 0 of Part 2.
8. Use of oral bisphosphonates following completion of Part 1 of the study.
9. Use of teriparatide or abaloparatide in the 2 months prior to Week 0 of Part 2.
10. Planned or recommended orthopedic surgery during the study.
11. History of traumatic fracture or orthopedic surgery within 6 months prior to Week 0 of Part 2.
12. Participants who are lactating.
13. Current active and symptomatic COVID-19 infection, or a history of suffering any long-term sequalae from COVID-19 infection.
14. Presence or history of any condition that, in the view of the investigator, places the participant at high risk of poor treatment compliance or of not completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2028-02-11 (Estimated); Study Completion 2028-05-10 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with TEAEs | For up to 44 weeks.
Part 1: Percentage of participants with TEAEs | For up to 44 weeks.
Part 2: Number of participants with TEAEs | For up to 52 weeks.
Part 2: Percentage of participants with TEAEs | For up to 52 weeks.
Part 1: Change from baseline for haematology laboratories values | For up to 44 weeks.
Part 2: Change from baseline for haematology laboratories values | For up to 52 weeks.
Part 1: Change from baseline for clinical chemistry laboratories values | For up to 44 weeks.
Part 2: Change from baseline for clinical chemistry laboratories values | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for FSH | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for FSH | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for estradiol | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for estradiol | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for temperature | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for temperature | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for pulse rate | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for pulse rate | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for respiratory rate | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for respiratory rate | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for systolic and diastolic blood pressure | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for systolic and diastolic blood pressure | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for QT | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for QT | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for QTc | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for QTc | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for QTCF | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for QTCF | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for QRS | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for QRS | For up to 52 weeks.
Part 1: Change from baseline in continuous variables for heart rate | For up to 44 weeks.
Part 2: Change from baseline in continuous variables for heart rate | For up to 52 weeks.
Part 1: The presence or absence of abnormality on ectopic mineralization, any sign of left ventricular hypertrophy or heart failures before and after administration of KK8123 on Echocardiogram | For up to 44 weeks.
Part 2: The presence or absence of abnormality on ectopic mineralization, any sign of left ventricular hypertrophy or heart failures before and after administration of KK8123 on Echocardiogram | For up to 52 weeks.
Part 1: Before and after administration presented at each time point in categorical variables for renal ultrasound | For up to 44 weeks.
Part 2: Before and after administration presented at each time point in categorical variables for renal ultrasound | For up to 52 weeks.
Part 1: KK8123 concentrations by maximum plasma concentration (Cmax) | For up to 44 weeks.
Part 2: KK8123 concentrations by maximum plasma concentration (Cmax) | For up to 52 weeks.
Part 1: KK8123 concentrations by maximum serum concentration (tmax) | For up to 44 weeks.
Part 2: KK8123 concentrations by maximum serum concentration (tmax) | For up to 52 weeks.
Part 1: KK8123 concentrations by area under the serum concentration time curve from zero to last detectable time point (AUClast) | For up to 44 weeks.
Part 2: KK8123 concentrations by area under the serum concentration time curve from zero to last detectable time point (AUClast) | For up to 52 weeks.
Part 1: KK8123 concentrations by the area under the serum concentration time curve from zero to infinity (AUC00-inf) | For up to 44 weeks.
Part 2: KK8123 concentrations by the area under the serum concentration time curve from zero to infinity (AUC00-inf) | For up to 52 weeks.
Part 1: KK8123 concentrations by apparent volume of distribution (V/F) | For up to 44 weeks..
Part 2: KK8123 concentrations by apparent volume of distribution (V/F) | For up to 52 weeks.
Part 1: KK8123 concentrations by terminal half-life (t1/2) | For up to 44 weeks.
Part 2: KK8123 concentrations by terminal half-life (t1/2) | For up to 52 weeks.
Part 1: KK8123 concentrations by apparent clearance (CL/F) | For up to 44 weeks.
Part 2: KK8123 concentrations by apparent clearance (CL/F) | For up to 52 weeks.
Part 1: KK8123 concentrations by maximum plasma concentration steady state (Cmax,ss) | For up to 44 weeks.
Part 2: KK8123 concentrations by maximum plasma concentration steady state (Cmax,ss) | For up to 52 weeks.
Part 1: KK8123 concentrations by time to maximum serum concentration steady state (tmax,ss) | For up to 44 weeks.
Part 2: KK8123 concentrations by time to maximum serum concentration steady state (tmax,ss) | For up to 52 weeks.
Part 1: KK8123 concentrations over time by area under the serum concentration curve within a dosing interval at steady state (AUCtau,ss) | For up to 44 weeks.
Part 2: KK8123 concentrations over time by area under the serum concentration curve within a dosing interval at steady state (AUCtau,ss) | For up to 52 weeks.
Part 1: KK8123 concentrations by time to steady state | For up to 44 weeks.
Part 2: KK8123 concentrations by time to steady state | For up to 52 weeks.
Part 1: KK8123 concentrations by accumulation ratio | For up to 44 weeks.
Part 2: KK8123 concentrations by accumulation ratio | For up to 52 weeks.
Part 1: To evaluate the effect of single and multiple SC administrations of KK8123 on serum phosphorus levels | For up to 44 weeks.
Part 2: To evaluate the effect of multiple SC administrations of KK8123 on serum phosphorus levels | For up to 52 weeks.

SECONDARY OUTCOMES:
Part 1: ADA positivity titers to be assessed by absolute number | For up to 44 weeks.
Part 1: ADA positivity titers to be assessed by percentage | For up to 44 weeks.
Part 2: ADA positivity titers to be assessed by absolute number | For up to 52 weeks.
Part 2: ADA positivity titers to be assessed by percentage | For up to 52 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kyowa Kirin, Study Chair — Kyowa Kirin, Inc.
Locations (9):
- United States (5):
  - University of California - San Francisco, San Francisco, California
  - Yale Center for XLH/ Yale University School of Medicine, New Haven, Connecticut
  - Indiana University School of Medicine University Hospital, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Hoptial Bictre, Le Kremlin-Bicêtre, Paris, France
- Germany (2):
  - Institute of Osteology and Biomechanics (IOBM), Hamburg
  - Universitaetsklinikum Wurzburg, Würzburg
- Hospital Universitario La Paz, Madrid, Spain